CLINICAL TRIAL: NCT03630575
Title: Study of Psychoactive Substances in Newborns' Hair Whose Mothers Were Treated and Followed at the Nice University Hospital - New Born Hair Study
Acronym: NBHS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigator never responded to requests for changes from the ethics committee.
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-PP-01
Record Dates: First submitted 2018-08-06; First posted 2018-08-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Newborns exposed in-utero to psychoactive substances (Experimental)
  Interventions: Procedure: Umbilical cord blood and hair collection

INTERVENTIONS:
Procedure: Umbilical cord blood and hair collection — At the birth of the newborn, a first hair sample and a cord blood sample will be taken. A follow-up of the newborn will be performed between 4 and 6 months in order to obtain a second hair sample.

SUMMARY:
Hair toxicological analysis is nowadays a complementary technique to blood and urinary analyses because it allows a better detection of xenobiotics in time.

The detection of xenobiotics is expressed in hours in blood and in days in urines; it is several months in the hair. So, hair makes it possible to establish a retrospective timetable of consumption and exposure to xenobiotics.

In newborns, hair has different morphological characteristics than adults' hair. It is thinner, more porous and the development phases are not the same.

Nevertheless, it is recognized that the absorption mechanisms of xenobiotics in newborns' hair are similar to those of adults. On the other hand, some difficulties of interpretation and discernment are observed between in utero exposure and environmental exposure after birth.

It is interesting to have data to estimate the absorption of psychoactive substances in newborns' hair following an utero exposure.

The main objective of this project is to study the mechanisms of incorporation of psychoactive substances administered to the mothers during pregnancy in newborns' hair.

ELIGIBILITY:
Inclusion Criteria:

* Newborns of mothers treated with known doses of psychoactive drugs during pregnancy or exposed to cannabinoids during pregnancy
* Full-term newborns (≥37 weeks)
* Informed consent signed by the child's legal representatives
* Affiliation to Social Security

Exclusion Criteria:

* Newborns of mothers exposed to unknown doses of psychoactive substances (excluding cannabis) during pregnancy
* One of the child's legal representatives hasn't signed the informed consent
* Premature delivery <37 weeks of amenorrhea
* Newborns who can't be followed at T 4-6 months.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Change of psychoactive substances concentration in newborn's hair at 6 months | At 6 Months
  The primary outcome measure is the presence of at least one molecule from the following classes of drugs (antidepressants, opioids, cannabinoids, anti-epileptics, benzodiazepines), on at least one of the hair segments studied, at a minimum concentration corresponding to the limit of quantification of the analytical technique.

CONTACTS AND LOCATIONS:
Overall Officials: André BONGAIN, PU-PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hôpital Archet 2 - Service de Gynécologie - Obstétrique - Reproduction, Nice, France